CLINICAL TRIAL: NCT04851756
Title: Immediate Effect of Capacitive Resistive Electric Transfer Therapy (CRet) Associated With Functional Massage on the Rectus Femoris and Gastrocnemius in Post-stroke Spasticity
Brief Title: Effects of CRet Associated With Functional Massage (F.M) on Gait and Functionality in Post-stroke Spasticity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Internacional de Catalunya (Other)
Responsible Party: Principal Investigator, Laura García Rueda, Principal Investigator, Universitat Internacional de Catalunya
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CRet2
Record Dates: First submitted 2021-04-11; First posted 2021-04-20 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Stroke Sequelae; Spasticity, Muscle; Massage; Electrotherapy
Keywords: Stroke; Spasticity; Functional Massage; CRet; Functionality; Gait
MeSH Terms: conditions — Muscle Spasticity; Stroke

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CRet Group (Experimental): 30 min CRet with F.M on the rectus femoris and gastrocnemius medialis and lateralis
  Interventions: Device: CRet
- CRet Sham Group (Sham Comparator): 30 min CRet with F.M on the rectus femoris and gastrocnemius medialis and lateralis with turned on CRet device at power 0
  Interventions: Device: Sham CRet

INTERVENTIONS:
Device: CRet — In prone position, subjects will get a 7 min preparation massage with CRet on resistive mode (80-100W), on the lumbar area, followed by a 5 min preparation massage with CRet on resistive mode (100-120 W) on the hamstrings. Then a 5 min Functional Massage (F.M) with passive anckle dorsiflexion and CRet on resistive mode (110-120 W) will be performed on the gastrocnemius medialis and lateralis, followed by a 4 min F.M with CRet on capacitive mode (180-250VA) on the mentioned area. In supine position, a 5 min F.M with passive knee flexion and CRet on resistive mode (110-140W) will be performed on the rectus femoris, followed by a 4 min F.M with passive knee flexion and CRet on capacitive mode (180-250VA) on the mentioned area. A physiotherapist will monitor the temperature of the patient's treated area every 2 minutes.
  Arms: CRet Group
Device: Sham CRet — In prone position, subjects will get a 7 min preparation massage with CRet on resistive mode (0 W), on the lumbar area, followed by a 5 min preparation massage with CRet on resistive mode (0 W) on the hamstrings. Then a 5 min Functional Massage (F.M) with passive anckle dorsiflexion and CRet on resistive mode (0 W) will be performed on the gastrocnemius medialis and lateralis, followed by a 4 min FM with CRet on capacitive mode (0 VA) on the mentioned area. In supine position, a 5 min F.M with passive knee flexion and CRet on resistive mode (0W) will be performed on the rectus femoris, followed by a 4 min F.M with passive knee flexion and CRet on capacitive mode (0VA) on the mentioned area.
  A physiotherapist will monitor the temperature of the patient's treated area every 2 minutes.
  Arms: CRet Sham Group

SUMMARY:
The purpose of this study is to assess the immediate effects of CRet associated to Functional Massage (F.M) in terms of gait and functionality after stroke

DETAILED DESCRIPTION:
Spasticity is a sensory motor disturbance as a result of a damage in the upper motoneuron, showing as an involuntary, intermittent and sustained activation of muscles. It is the most common feature after stroke, which most affects motor and functional recovery.

Spasticity prevalence runs from 25% to 46% after the first six months post-stroke, and it is estimated that 16% will require treatment.

Spasticity has neural (increased reflex activity) and biomechanical (altered viscoelastic properties due to immobilization) components. The initial paralysis after stroke modifies the bio mechanical properties of the muscle, thus shortening its fibers and causing an increase of velocity-dependent reflexes in the affected area. Spasticity manifests with paresis, increased muscle tone, muscular hyperactivity, decreased range of movement and pain.

Gait disorder is one of the main physical limitations in stroke survivors and an important target for stroke rehabilitation, since physiotherapy treatments of spasticity aim to decrease excessive muscular tone, ease mobility, give the patient the sense of right position and avoid joint limitations.

Functional Massage (F.M) is a non-invasive manual therapy technique that combines rhythmical passive mobilizations of the joints with gentle massage and compression of the muscles to be treated. As massage therapy is effective to improve spastic muscles and gross motor functions, F.M may be appropriate in treating post stroke spasticity and gait function. No studies were found on its effectiveness in patients with post-stroke spasticity.

Capacitive Resistive electric transfer therapy (CRet) is a non-invasive diathermy technique that, providing high frequency energy (300KHz-1.2MHz),generates a thermal effect on soft tissues. CRet is used to facilitate tissue regeneration, and it does not need a surface-cooling system as its wave frequency is lower than in conservative diathermy. Its effectiveness has been evaluated in several studies related to musculoskeletal disorders, where an increase in temperature is needed in deep tissues in order to generate changes on its viscoelasticity.

This effect may be beneficial in the spasticity treatment since spasticity onset and development may be affected by structural changes in muscular and tendinous fibers, as well as in its intra and extracellular components.

No studies on the effects of CRet in post-stroke spasticity treatment were found.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of stroke
* Scoring 1+ on the Modified Ashworth Scale (MAS) for hip flexion and/or knee flexion or/and ancke dorsiflexion on the most affected limb
* Scoring 25 or plus on the Montreal Cognitive Assessment (MoCA)
* Signing the informed consent form

Exclusion Criteria:

* Having suffered a traumatism on the lower limbs three months, or less, before the intervention
* Other neurological diseases
* Presence of osteosynthetic material
* Pacemaker wearing
* Treatment with botulinum toxin or another antispastic medication, six months , or less, before the intervention
* Carry baclofen pump
* Functional inability to adopt the prone or supine position on the treatment table
* Functional inability to sit, stand and walk
* Poor language and communication skills that make difficult to understand the informed consent form
* Contraindications to Functional Massage (infectious diseases, inflammatory vascular conditions, acute inflammation, haemorrhagia, fever)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2021-04-29 (Actual); Primary Completion 2022-05-27 (Actual); Study Completion 2022-09-05 (Actual)

PRIMARY OUTCOMES:
Gait Performance | T1: Baseline, T2: Immediately after treatment and T3: follow up 30 minutes after treatment ]
  To evaluate change in gait speed after one session with CRet associated to F.M by the 4-metre-walk-test (4MWT). The assessor will indicate the participant to walk 4m at her fastest velocity. The timing will ve recorded.
Functional Lower Extremity Force | T1: Baseline, T2: Immediately after treatment and T3: follow up 30 minutes after treatment ]
  To evaluate change in functional lower extremity force after one session with CRet associated to F.M by the 5 times sit-to-stand test. Participants will be in the seating position on the treatment bed, and will stand and sit for five times. Time will start when the tester says 'go'.Time will stop when the participant's body touches the chair following the fifth repetition.

SECONDARY OUTCOMES:
Active Range of Movement (AROM) of the anckle | T1: Baseline, T2: Immediately after treatment and T3: follow up 30 minutes after treatment ]
  Measuring change of the maximum range of active dorsiflexion with an inclinometer by the dorsiflexion lunge test. The participant will be standing and holding on a wall. The tester will ask the participant to bend her ankle to her maximum range without lifting her heel from the floor.
AROM of the knee | T1: Baseline, T2: Immediately after treatment and T3: follow up 30 minutes after treatment ]
  Measuring change of the maximum range of active knee flexion on three point ( 0= no knee flexion, 1= knee does not reach = or < 90 degrees, 2= knee flexion >90 ) Fugl Meyer Assessment. Only the lower extremity item of the Fugl Meyer assessment will be used in this study.
Global Improvement | Baseline up 30 min after treatment
  Global Improvement on two 5 points Likert Scale questions:
  (1) Strongly disagree; (2) Disagree; (3) Neither agree nor disagree; (4) Agree; (5) Strongly agree.

CONTACTS AND LOCATIONS:
Overall Officials: Rosa Cabanas-Valdés, PhD, Principal Investigator — Universitat Internacional de Catalunya
Locations (1):
- Assessment Room at UIC Sant Cugat, Sant Cugat del Vallès, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pandyan AD, Gregoric M, Barnes MP, Wood D, Van Wijck F, Burridge J, Hermens H, Johnson GR. Spasticity: clinical perceptions, neurological realities and meaningful measurement. Disabil Rehabil. 2005 Jan 7-21;27(1-2):2-6. doi: 10.1080/09638280400014576. No abstract available. PMID 15799140
- [Background] Zorowitz RD, Gillard PJ, Brainin M. Poststroke spasticity: sequelae and burden on stroke survivors and caregivers. Neurology. 2013 Jan 15;80(3 Suppl 2):S45-52. doi: 10.1212/WNL.0b013e3182764c86. PMID 23319485
- [Background] Sainz-Pelayo MP, Albu S, Murillo N, Benito-Penalva J. [Spasticity in neurological pathologies. An update on the pathophysiological mechanisms, advances in diagnosis and treatment]. Rev Neurol. 2020 Jun 16;70(12):453-460. doi: 10.33588/rn.7012.2019474. Spanish. PMID 32500524
- [Background] Wissel J, Verrier M, Simpson DM, Charles D, Guinto P, Papapetropoulos S, Sunnerhagen KS. Post-stroke spasticity: predictors of early development and considerations for therapeutic intervention. PM R. 2015 Jan;7(1):60-7. doi: 10.1016/j.pmrj.2014.08.946. Epub 2014 Aug 27. PMID 25171879
- [Background] Gracies JM. Pathophysiology of spastic paresis. I: Paresis and soft tissue changes. Muscle Nerve. 2005 May;31(5):535-51. doi: 10.1002/mus.20284. PMID 15714510
- [Background] Gracies JM. Pathophysiology of spastic paresis. II: Emergence of muscle overactivity. Muscle Nerve. 2005 May;31(5):552-71. doi: 10.1002/mus.20285. PMID 15714511
- [Background] Wang Y, Mukaino M, Ohtsuka K, Otaka Y, Tanikawa H, Matsuda F, Tsuchiyama K, Yamada J, Saitoh E. Gait characteristics of post-stroke hemiparetic patients with different walking speeds. Int J Rehabil Res. 2020 Mar;43(1):69-75. doi: 10.1097/MRR.0000000000000391. PMID 31855899
- [Background] Tricás JM. Cuadernillos Prácticos de Fisioterapia, Masaje Funcional. Zaragoza: Fundación Empresa Universidad de Zaragoza. 2001;4.
- [Background] Barra-López M.E, Castillo-Tomás S, González-Rueda V, Villar-Mateo E, N. Domene- Guinart N y López-de-Celis C. Efectividad del masaje funcional en el síndrome de impingement subacromial. Fisioterapia 2015; 37 (2): 75
- [Background] Clijsen R, Leoni D, Schneebeli A, Cescon C, Soldini E, Li L, Barbero M. Does the Application of Tecar Therapy Affect Temperature and Perfusion of Skin and Muscle Microcirculation? A Pilot Feasibility Study on Healthy Subjects. J Altern Complement Med. 2020 Feb;26(2):147-153. doi: 10.1089/acm.2019.0165. Epub 2019 Oct 3. PMID 31580698
- [Background] Lopez-de-Celis C, Hidalgo-Garcia C, Perez-Bellmunt A, Fanlo-Mazas P, Gonzalez-Rueda V, Tricas-Moreno JM, Ortiz S, Rodriguez-Sanz J. Thermal and non-thermal effects off capacitive-resistive electric transfer application on the Achilles tendon and musculotendinous junction of the gastrocnemius muscle: a cadaveric study. BMC Musculoskelet Disord. 2020 Jan 20;21(1):46. doi: 10.1186/s12891-020-3072-4. PMID 31959172
- [Background] H. Bingöl, Ö. Yılmaz. Effects of functional massage on spasticity and motor functions in children with cerebral palsy: a randomized controlled study. Journal of Exercise Therapy and Rehabilitation. 2018; 5:135-142.
- [Background] Yokota, Y., Tashiro, Y., Suzuki, Y., Tasaka, S., et al. (2017). Effect of capacitive and resistive electric transfer on tissue temperature, muscle flexibility, and blood circulation. J. Nov. Physiother. 7:325.
- [Background] Osti R, Pari C, Salvatori G, Massari L. Tri-length laser therapy associated to tecar therapy in the treatment of low-back pain in adults: a preliminary report of a prospective case series. Lasers Med Sci. 2015 Jan;30(1):407-12. doi: 10.1007/s10103-014-1684-3. Epub 2014 Nov 7. PMID 25376670
- [Background] Coccetta CA, Sale P, Ferrara PE, Specchia A, Maccauro G, Ferriero G, Ronconi G. Effects of capacitive and resistive electric transfer therapy in patients with knee osteoarthritis: a randomized controlled trial. Int J Rehabil Res. 2019 Jun;42(2):106-111. doi: 10.1097/MRR.0000000000000324. PMID 30362981
- [Background] Rikli R, Jones C, Functional fitness normative scores for community-residing older adults, ages 60-94. J Aging Phys Activity 1999;7(2):162-81.
- [Background] Bloem AEM, Veltkamp M, Spruit MA, Custers JWH, Bakker EWP, Dolk HM, Grutters JC. Validation of 4-meter-gait-speed test and 5-repetitions-sit-to-stand test in patients with pulmonary fibrosis: a clinimetric validation study. Sarcoidosis Vasc Diffuse Lung Dis. 2018;35(4):317-326. doi: 10.36141/svdld.v35i4.7035. Epub 2020 Mar 9. PMID 32476919
- [Background] Scrivener K, Schurr K, Sherrington C. Responsiveness of the ten-metre walk test, Step Test and Motor Assessment Scale in inpatient care after stroke. BMC Neurol. 2014 Jun 16;14:129. doi: 10.1186/1471-2377-14-129. PMID 24934859
- [Background] Clanton TO, Matheny LM, Jarvis HC, Jeronimus AB. Return to play in athletes following ankle injuries. Sports Health. 2012 Nov;4(6):471-4. doi: 10.1177/1941738112463347. PMID 24179584
- [Background] Dobkin BH, Firestine A, West M, Saremi K, Woods R. Ankle dorsiflexion as an fMRI paradigm to assay motor control for walking during rehabilitation. Neuroimage. 2004 Sep;23(1):370-81. doi: 10.1016/j.neuroimage.2004.06.008. PMID 15325385
- [Background] Rech KD, Salazar AP, Marchese RR, Schifino G, Cimolin V, Pagnussat AS. Fugl-Meyer Assessment Scores Are Related With Kinematic Measures in People with Chronic Hemiparesis after Stroke. J Stroke Cerebrovasc Dis. 2020 Jan;29(1):104463. doi: 10.1016/j.jstrokecerebrovasdis.2019.104463. Epub 2019 Nov 15. PMID 31740027
- [Background] Perez-Bellmunt A, Simon M, Lopez-de-Celis C, Ortiz-Miguel S, Gonzalez-Rueda V, Fernandez-de-Las-Penas C. Effects on Neuromuscular Function After Ischemic Compression in Latent Trigger Points in the Gastrocnemius Muscles: A Randomized Within-Participant Clinical Trial. J Manipulative Physiol Ther. 2022 Sep;45(7):490-496. doi: 10.1016/j.jmpt.2020.07.015. Epub 2021 Jan 9. PMID 33431281